CLINICAL TRIAL: NCT04811482
Title: A Pilot Study of a School-Based Treatment for Early Childhood Anxiety
Brief Title: School-Based Treatment for Early Childhood Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-2523
Record Dates: First submitted 2021-03-18; First posted 2021-03-23 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Anxiety
Keywords: Parent-Child Interaction Therapy (PCIT); CALM Protocol; Teacher-Child Interaction Training (TCIT)
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is a pilot study in which all individuals will be enrolled in the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): This study consists of one arm, an intervention group.
  Interventions: Behavioral: TCIT-CALM (Teacher-Child Interaction Training-CALM)

INTERVENTIONS:
Behavioral: TCIT-CALM (Teacher-Child Interaction Training-CALM) — This intervention is designed to treat early childhood anxiety. It is an adaptation of parent-child interaction therapy (PCIT), in which teachers rather than parents are targeted as the therapeutic agent of change. The intervention follows the procedures of the CALM protocol, in which caregivers are taught play therapy skills to support and address anxious behaviors and avoidance.

SUMMARY:
This pilot will be used for academic research, in hopes of developing effective treatments for early childhood anxiety. The intervention is an adaptation of Parent-Child Interaction Therapy (PCIT). PCIT is an evidence-based intervention, rooted in attachment and social learning theory. In recent years, researchers have successfully adapted PCIT to address anxiety in a clinical setting (PCIT-CALM). In this pilot study, we will be applying the PCIT-CALM intervention in the school setting, emphasizing teachers as a therapeutic agent of change.

PCIT is unique because the child's caregiver is trained on how to use therapeutic techniques, and then receives live coaching via a "bug in the ear" as they learn to implement the new skills. In this pilot study, both parents and teachers will be taught skills to create a therapeutic relationship and address anxiety. After these teaching sessions, the child's teacher will receive coaching in the classroom to implement the skills. The intervention will last approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Scores in the at-risk or clinical range for anxiety on the BASC-3 or CBCL (which will be filled out by a parent and teacher to determine eligibility)
* Child must be enrolled at the Montessori School of Denver where the intervention is being conducted.

Exclusion Criteria:

* None if other criteria are met.
* Comorbidity will not exclude a child, but if comorbidities are discovered for which there are other evidence-based treatments available, parents will be encouraged to seek additional resources.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Measuring Changes in scores on Behavior Assessment System for Children (BASC-3) | Pre- treatment Baseline and immediately following the intervention; An additional data collection was later added for longitudinal data that will be collected in October.
  A normed clinical rating scale for assessing behavior and mental health; This tool was chosen due to the norms for young children and the ability to have both parent and teacher rating scales.
Measuring Changes in scores on Child Behavior Checklist (CBCL) | Pre- treatment Baseline and immediately following the intervention; An additional data collection was later added for longitudinal data that will be collected in October.
  A normed clinical rating scale for assessing behavior and mental health; This tool was chosen due to the norms for young children and the ability to have both parent and teacher rating scales.

SECONDARY OUTCOMES:
Therapy Attitude Inventory | Immediately following the intervention
  A brief questionnaire to assess how well the intervention worked for the adults involved. The questionnaire includes 10 questions with a Likert scale response (1-5; 1 indicating little value from the intervention and 5 indicating it was highly beneficial.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Virlee, Principal Investigator — University of Colorado, Denver
Locations (1):
- Montessori School of Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
Currently, there is no plan to share IPD, but if data would be useful to others it has not been ruled out.

REFERENCES:
- [Background] Puliafico, A. C., Furr, J. M., Hong, N, & Comer, J. S. (2020). The CALM program for early childhood anxiety: Version 2.0.
- [Background] Puliafico AC, Comer JS, Pincus DB. Adapting parent-child interaction therapy to treat anxiety disorders in young children. Child Adolesc Psychiatr Clin N Am. 2012 Jul;21(3):607-19. doi: 10.1016/j.chc.2012.05.005. Epub 2012 Jun 2. PMID 22800997
- [Background] Comer JS, Puliafico AC, Aschenbrand SG, McKnight K, Robin JA, Goldfine ME, Albano AM. A pilot feasibility evaluation of the CALM Program for anxiety disorders in early childhood. J Anxiety Disord. 2012 Jan;26(1):40-9. doi: 10.1016/j.janxdis.2011.08.011. Epub 2011 Aug 25. PMID 21917417